CLINICAL TRIAL: NCT06094829
Title: Tobacco and Alcohol Influence on Oncogenic Drivers and Somatic Evolution in the Oral Mucosa
Acronym: DEMO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0749
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Oral cytobrush; Healthy oral mucosa; Oral squamous cell carcinoma; Tobacco and alcohol
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Oral cytobrush samples will be collected (1 per patient, single time point without follow-up) and analysed via deep whole exome sequencing (>500x).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers: Healthy subjects having smoked 100 cigarettes or more during their life.
  Interventions: Other: Oral cytobrush
- Non-smokers: Healthy subjects having smoked less than 100 cigarettes during their life.
  Interventions: Other: Oral cytobrush

INTERVENTIONS:
Other: Oral cytobrush — Oral epithelial cells will be collected during routine odontology appointments, upon documented non-opposition, via minimally invasive cytobrush sampling of the inner cheek

SUMMARY:
Head and neck cancers represent more than 500,000 cases per year worldwide, and often involve post-treatment relapse. The oral cavity is the most frequent site, but early disease stages are still insufficiently characterised and poorly detected. The study's aim is to better understand the oral mucosa somatic evolution, and how it can give rise to oral squamous cell carcinoma (OSCC).

This is a multi-centric, descriptive, non-interventional cohort in healthy adult subjects. The aim of the study is to detect the presence of OSCC driver gene mutations in healthy subjects' oral mucosa, quantify whether they provide cells with a selective advantage, and study the impact of tobacco and alcohol consumption on the mutational load. This study will not allow to identify potential malignant cells, and will be usable for diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 or more.
* Subject coming to odontology practice for routine visit.
* Subject having accepted to participate to the research by oral non-opposition
* Subject having given additional written consent for genetic studies.
* Smoking group criterion: subjects having smoked 100+ cigarettes/joints during their life.

Exclusion Criteria:

* Personal history of cancer, whichever the type.
* Treatment with anticoagulants or platelet aggregation inhibitors.
* Bilateral lesions of the inner cheek preventing painless biological sample collection.
* Subject under under guardians or curators
* Pregnancy or breastfeeding
* Cannabis usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects coming to odontology practices for routine visits
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of non-synonymous OSCC driver mutations in the healthy mucosa of smokers | 12 months
  Difference in mean number of non-synonymous mutations found in OSCC driver genes between smokers and non-smokers.

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Cabinet Libéral Picquendar, Bougival
  - Cabinet Libéral Balayre, Chassieu
  - Cabinet Libéral Debeauvais, Châtillon-Coligny
  - Cabinet Libéral Finet, Fontaine-lès-Dijon
  - Cabinet Libéral Jaeggy, Haguenau
  - Unité de chirurgie et médecine orales (UCMO) - HCL - Hôpital Edouard Herriot- Pavillon R, Lyon
  - Centre de Consultations et de Traitements Dentaires HCL, Lyon
  - Cabinet Libéral Grammatica, Lyon
  - Cabinet Libéral Cougot, Meudon
  - Cabinet Libéral Calvo, Quint-Fonsegrives
  - Cabinet Libéral Glomet, Saumur
  - Cabinet Libéral Dutour, Theix
  - Cabinet Libéral Masri, Vandœuvre-lès-Nancy
  - Cabinet Libéral Bondil, Villefranche-sur-Saône
  - Cabinet Libéral Janisset-Masse, Villiers-sur-Marne